CLINICAL TRIAL: NCT02761330
Title: Cognitive Recovery After Electroconvulsive Therapy and General Anesthesia Reconstitution of Consciousness and Cognition (Phase 2)
Brief Title: Cognitive Recovery After Electroconvulsive Therapy and General Anesthesia
Acronym: RCC2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: James S McDonnell Foundation (Other)
Responsible Party: Principal Investigator, Ben Palanca, Assistant Professor of Anesthesiology, Washington University School of Medicine
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 201512110
Record Dates: First submitted 2016-04-30; First posted 2016-05-04 (Estimated); Results first posted 2021-06-28 (Actual); Last update posted 2021-06-28 (Actual); Status verified 2021-06

CONDITIONS: Depression; Delirium; Seizures; Cognitive Disorders
Keywords: Anesthesia; Electroconvulsive therapy; Delirium; Electroencephalography; Seizures; Depression; Ketamine; Etomidate; Physiological Effects of Drugs; Pharmacologic Actions; Confusion; Mental Disorders; Neurobehavioral Manifestations; Signs and Symptoms; Neurologic Manifestations; Cognitive Disorders
MeSH Terms: conditions — Depression; Delirium; Seizures; Cognitive Dysfunction; Confusion; Mental Disorders; Neurobehavioral Manifestations; Signs and Symptoms; Neurologic Manifestations | interventions — Ketamine; Electroconvulsive Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Etomidate + ECT (Active Comparator): General anesthesia for ECT will be induced with etomidate, approximately 0.2 mg/kg (0.1-0.6 mg/kg). Following application of stimulation electrodes to the patients scalp, an ECT charge will be administered at the previously determined therapeutic dose.
  Interventions: Procedure: Electroconvulsive Therapy
- Ketamine + ECT (Experimental): General anesthesia for ECT will be induced with ketamine, approximately 2 mg/kg (1-2.5 mg/kg). Following application of stimulation electrodes to the patients scalp, an ECT charge will be administered at the previously determined therapeutic dose.
  Interventions: Drug: Ketamine; Procedure: Electroconvulsive Therapy
- Ketamine alone (Sham Comparator): General anesthesia for ECT will be induced with ketamine, approximately 2 mg/kg (1-2.5 mg/kg). Following application of stimulation electrodes to the patients scalp, no ECT charge will be administered.
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Ketamine — Ketamine will be used to induce general anesthesia with or without subsequent ECT. Within a single patient, the dose will remain consistent throughout the study and is estimated to be 2 mg/kg.
  Arms: Ketamine + ECT; Ketamine alone
Procedure: Electroconvulsive Therapy — Dose of the ECT charge will be determined during titration session prior to randomization.
  Other Names: ECT
  Arms: Etomidate + ECT; Ketamine + ECT

SUMMARY:
This study is geared toward characterizing the recovery of brain activity and cognitive function following treatments of electroconvulsive therapy and ketamine general anesthesia.

DETAILED DESCRIPTION:
Seizures are often associated with loss of consciousness, possibly through effects on sub-cortical arousal systems, disruption of cortical-subcortical interactions, and ultimately through depressed neocortical function. Furthermore, people are often confused in the post-ictal state even when consciousness returns after a seizure. Disrupted cognitive function during the postictal phase has not been fully characterized but presents short and long-term implications. Many experience an acute disorder of attention, consciousness, and cognition, referred to as delirium. Memory deficits are also common. The neurobiology for these phenomena are incomplete and challenging to test, as seizures are typically sporadic and vary in intensity and character. In contrast, the setting of electroconvulsive therapy (ECT) provides the opportunity to study the reconstitution of consciousness and cognition following seizures in an elective and predictable context.

There is no standard agent used to induce general anesthesia during ECT. Ketamine is receiving greater attention as an infusion for treating depression and for its potential benefits on improving ECT efficacy and expediting cognitive recovery. Further data are needed to determine whether ketamine may improve recovery of cognitive function relative to etomidate, a commonly used anesthetic for general anesthesia during ECT.

The investigators will evaluate the cognition function and electroencephalographic patterns that accompany the recovery from ECT and general anesthesia. Twenty patients with refractory depression will be randomized in this interventional single-blinded randomized crossover trial. Each patient will complete seven study visits. The first visit will be conducted during the dose-charge titration ECT treatment with etomidate anesthesia. After this session, patients will be randomized to three sessions each week for two weeks (six treatments total). Over the first week patients will be randomized in order for three treatment arms: (1) etomidate general anesthesia and ECT, (2) ketamine general anesthesia and ECT, and (3) ketamine alone. Patients will be blinded to the treatment arm for each session. Baseline and post-treatment measurements of cognition and ECT will be acquired on each of the six treatment sessions.

Patients that agree will have a MRI.

ELIGIBILITY:
Inclusion Criteria:

* Treatment resistant depression requiring outpatient ECT
* Planned right unilateral ECT stimulation
* English speaking
* Able to provide written informed consent

Exclusion Criteria:

* Known brain lesion or neurological illness that causes cognitive impairment
* Schizophrenia
* Schizoaffective disorder
* Blindness or deafness or motor impediments that may impair performance for cognitive testing battery
* Inadequate ECT seizure duration with etomidate

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2019-09-11 (Actual); Study Completion 2019-09-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hickman LB, Kafashan M, Labonte AK, Chan CW, Huels ER, Guay CS, Guan MJ, Ching S, Lenze EJ, Farber NB, Avidan MS, Hogan RE, Palanca BJA. Postictal generalized electroencephalographic suppression following electroconvulsive therapy: Temporal characteristics and impact of anesthetic regimen. Clin Neurophysiol. 2021 Apr;132(4):977-983. doi: 10.1016/j.clinph.2020.12.018. Epub 2021 Jan 28. PMID 33652270
- [Derived] Hickman LB, Hogan RE, Labonte AK, Kafashan M, Chan CW, Huels ER, Ching S, Lenze EJ, Maccotta L, Eisenman LN, Keith Day B, Farber NB, Avidan MS, Palanca BJA. Voltage-based automated detection of postictal generalized electroencephalographic suppression: Algorithm development and validation. Clin Neurophysiol. 2020 Dec;131(12):2817-2825. doi: 10.1016/j.clinph.2020.08.015. Epub 2020 Sep 11. PMID 33137572
- [Derived] Palanca BJA, Maybrier HR, Mickle AM, Farber NB, Hogan RE, Trammel ER, Spencer JW, Bohnenkamp DD, Wildes TS, Ching S, Lenze E, Basner M, Kelz MB, Avidan MS. Cognitive and Neurophysiological Recovery Following Electroconvulsive Therapy: A Study Protocol. Front Psychiatry. 2018 May 14;9:171. doi: 10.3389/fpsyt.2018.00171. eCollection 2018. PMID 29867602

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 17 patients were enrolled for study participation between May 2016 and July 2018 at Barnes Jewish Hospital in St. Louis, MO.
Pre-assignment Details: 14 of 17 participants were randomized. Of those not randomized, 1 participant's treatment course was canceled by clinical staff, 1 participant withdrew consent prior to any study participation, and 1 participant was deemed ineligible.
Groups:
- Ketamine +ECT, Etomidate + ECT, Ketamine Sham: Participants first received ECT treatment under Ketamine general anesthesia, then ECT treatment under Etomidate anesthesia, and finally participants received Ketamine general anesthesia with sham ECT.
  Ketamine+ECT: General anesthesia for ECT will be induced with ketamine, approximately 2 mg/kg (1-2.5 mg/kg). Following application of stimulation electrodes to the patients scalp, an ECT charge will be administered at the previously determined therapeutic dose.
  Ketamine Sham: General anesthesia for ECT will be induced with ketamine, approximately 2 mg/kg (1-2.5 mg/kg). Following application of stimulation electrodes to the patients scalp, no ECT charge will be administered.
  Etomidate + ECT: General anesthesia for ECT will be induced with etomidate, approximately 0.2 mg/kg (0.1-0.6 mg/kg). Following application of stimulation electrodes to the patients scalp, an ECT charge will be administered at the previously determined therapeutic dose.
- Ketamine +ECT, Ketamine Sham, Etomidate + ECT: Participants first received ECT treatment under Ketamine general anesthesia, then Ketamine general anesthesia with sham ECT and finally participants received ECT treatment under Etomidate anesthesia.
  Ketamine+ECT: General anesthesia for ECT will be induced with ketamine, approximately 2 mg/kg (1-2.5 mg/kg). Following application of stimulation electrodes to the patients scalp, an ECT charge will be administered at the previously determined therapeutic dose.
  Ketamine Sham: General anesthesia for ECT will be induced with ketamine, approximately 2 mg/kg (1-2.5 mg/kg). Following application of stimulation electrodes to the patients scalp, no ECT charge will be administered.
  Etomidate + ECT: General anesthesia for ECT will be induced with etomidate, approximately 0.2 mg/kg (0.1-0.6 mg/kg). Following application of stimulation electrodes to the patients scalp, an ECT charge will be administered at the previously determined therapeutic dose.
- Etomidate +ECT, Ketamine + ECT, Ketamine Sham: Participants first received ECT treatment under Etomidate general anesthesia, then ECT treatment under Ketamine general anesthesia and finally participants received Ketamine general anesthesia with sham ECT.
  Ketamine+ECT: General anesthesia for ECT will be induced with ketamine, approximately 2 mg/kg (1-2.5 mg/kg). Following application of stimulation electrodes to the patients scalp, an ECT charge will be administered at the previously determined therapeutic dose.
  Ketamine Sham: General anesthesia for ECT will be induced with ketamine, approximately 2 mg/kg (1-2.5 mg/kg). Following application of stimulation electrodes to the patients scalp, no ECT charge will be administered.
  Etomidate + ECT: General anesthesia for ECT will be induced with etomidate, approximately 0.2 mg/kg (0.1-0.6 mg/kg). Following application of stimulation electrodes to the patients scalp, an ECT charge will be administered at the previously determined therapeutic dose.
- Etomidate +ECT, Ketamine Sham, Ketamine +ECT: Participants first received ECT treatment under Etomidate general anesthesia, then Ketamine general anesthesia with sham ECT and finally participants received ECT treatment under Ketamine anesthesia.
  Ketamine+ECT: General anesthesia for ECT will be induced with ketamine, approximately 2 mg/kg (1-2.5 mg/kg). Following application of stimulation electrodes to the patients scalp, an ECT charge will be administered at the previously determined therapeutic dose.
  Ketamine Sham: General anesthesia for ECT will be induced with ketamine, approximately 2 mg/kg (1-2.5 mg/kg). Following application of stimulation electrodes to the patients scalp, no ECT charge will be administered.
  Etomidate + ECT: General anesthesia for ECT will be induced with etomidate, approximately 0.2 mg/kg (0.1-0.6 mg/kg). Following application of stimulation electrodes to the patients scalp, an ECT charge will be administered at the previously determined therapeutic dose.
- Ketamine Sham, Etomidate +ECT, Ketamine +ECT: Participants first received Ketamine general anesthesia with sham ECT, then ECT treatment under Etomidate general anesthesia and finally participants received ECT treatment under Ketamine anesthesia.
  Ketamine+ECT: General anesthesia for ECT will be induced with ketamine, approximately 2 mg/kg (1-2.5 mg/kg). Following application of stimulation electrodes to the patients scalp, an ECT charge will be administered at the previously determined therapeutic dose.
  Ketamine Sham: General anesthesia for ECT will be induced with ketamine, approximately 2 mg/kg (1-2.5 mg/kg). Following application of stimulation electrodes to the patients scalp, no ECT charge will be administered.
  Etomidate + ECT: General anesthesia for ECT will be induced with etomidate, approximately 0.2 mg/kg (0.1-0.6 mg/kg). Following application of stimulation electrodes to the patients scalp, an ECT charge will be administered at the previously determined therapeutic dose.
- Ketamine Sham, Ketamine +ECT, Etomidate +ECT: Participants first received Ketamine general anesthesia with sham ECT, then ECT treatment under Ketamine general anesthesia and finally participants received ECT treatment under Etomidate anesthesia.
  Ketamine+ECT: General anesthesia for ECT will be induced with ketamine, approximately 2 mg/kg (1-2.5 mg/kg). Following application of stimulation electrodes to the patients scalp, an ECT charge will be administered at the previously determined therapeutic dose.
  Ketamine Sham: General anesthesia for ECT will be induced with ketamine, approximately 2 mg/kg (1-2.5 mg/kg). Following application of stimulation electrodes to the patients scalp, no ECT charge will be administered.
  Etomidate + ECT: General anesthesia for ECT will be induced with etomidate, approximately 0.2 mg/kg (0.1-0.6 mg/kg). Following application of stimulation electrodes to the patients scalp, an ECT charge will be administered at the previously determined therapeutic dose.
Period: Treatment Week 1
Arm/Group | Ketamine +ECT, Etomidate + ECT, Ketamine Sham | Ketamine +ECT, Ketamine Sham, Etomidate + ECT | Etomidate +ECT, Ketamine + ECT, Ketamine Sham | Etomidate +ECT, Ketamine Sham, Ketamine +ECT | Ketamine Sham, Etomidate +ECT, Ketamine +ECT | Ketamine Sham, Ketamine +ECT, Etomidate +ECT
Started | 2 | 3 | 2 | 3 | 1 | 3
Completed | 2 | 3 | 2 | 2 | 1 | 2
Not Completed | 0 | 0 | 0 | 1 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0 | 1
Period: Treatment Week 2
Arm/Group | Ketamine +ECT, Etomidate + ECT, Ketamine Sham | Ketamine +ECT, Ketamine Sham, Etomidate + ECT | Etomidate +ECT, Ketamine + ECT, Ketamine Sham | Etomidate +ECT, Ketamine Sham, Ketamine +ECT | Ketamine Sham, Etomidate +ECT, Ketamine +ECT | Ketamine Sham, Ketamine +ECT, Etomidate +ECT
Started | 2 | 3 | 2 | 1 (1 pt. in this group completed Week 1, but did not begin Week 2 due to withdraw.) | 1 | 1 (1 pt. in this group completed Week 1, but did not begin Week 2 due to cancellation of treatment.)
Completed | 2 | 3 | 2 | 1 | 1 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Per the participant flow report, 17 patients were enrolled in study procedures. Only 10 completed the study, per the full protocol, as reported. However, data from 15 participants are eligible for analyses. So, all analyses were done with 15 participants.
Groups:
- AllParticipants: All participants enrolled in study procedures.
Arm/Group | AllParticipants
Number analyzed (Participants) | 15
Age, Continuous [Median (Standard Deviation); unit: years] | 37 (13.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 15
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 15
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Cognitive Function During Recovery: Rate of Recovery
Description: A cognitive test battery was administered at 0, 30, 60, 90, and 120 minutes following return of consciousness after general anesthesia on each treatment day (1-6). The data from each treatment day (1-6) were averaged for analyses.
  Cognition Test Battery:
  * Psychomotor Vigilance Task (PVT)
  * Digital Symbol Substitution Task (DSST)
  * Motor Praxis Task (MP)
  * Visual Object Learning Task (VOLT)
  * Abstract Matching (AM)
  Rate of Recovery for this measure is defined as the time (in inverse hours) for participants to return to their baseline performance for each task.
Time Frame: 0, 30, 60, 90, 120 minutes following return of consciousness, assessed on treatment days 1-6.
Population: Participants with cogntive task data complete for the majority of timepoints following return of responsiveness for more than one treatment day were included in analyses. Additional participants were excluded for individual cognitive task measures for being extreme outliers.
Measure: Median (Inter-Quartile Range); unit: inverse hours
Arm/Group | Etomidate + ECT | Ketamine + ECT | Ketamine Alone
Number analyzed (Participants) | 9 | 9 | 11
inverse hours
  PVT Reaction Time: number analyzed (Participants) | 7 | 9 | 11
  PVT Reaction Time | 3.5 [2.2 to 4.0] | 6.3 [5.4 to 7.1] | 24.7 [8.1 to 27.5]
  DSST Reaction Time: number analyzed (Participants) | 8 | 9 | 11
  DSST Reaction Time | 9.7 [6.8 to 10] | 3.0 [2.2 to 3.1] | 2.9 [2.4 to 3.7]
  MP Reaction Time | 3.9 [3.5 to 4.4] | 2.5 [1.4 to 3.1] | 2.6 [2.6 to 2.6]
  VOLT Reaction Time: number analyzed (Participants) | 9 | 7 | 11
  VOLT Reaction Time | 9.2 [8.9 to 9.3] | 11.6 [5.2 to 12.8] | 3.1 [2.8 to 3.3]
  AM Reaction Time | 4.8 [4.8 to 4.8] | 1.6 [1.6 to 1.6] | 2.3 [2.2 to 2.4]
Statistical Analysis 1: Comparison: Etomidate + ECT vs Ketamine + ECT; Comparison between the Etomidate + ECT and Ketamine + ECT groups for the recovery rate of Psychomotor Vigilance Task (PVT) reaction time; Test type: Other; p = 0.016, Wilcoxon Signed-Ranked Test — Not adjusted for multiple comparisons
Statistical Analysis 2: Comparison: Ketamine + ECT vs Ketamine Alone; Comparison between the Ketamine + ECT and Ketamine Alone groups for the recovery rate of Psychomotor Vigilance Task (PVT) reaction time; Test type: Other; p = 0.012, Wilcoxon Signed-Ranked Test — Not adjusted for multiple comparisons
Statistical Analysis 3: Comparison: Etomidate + ECT vs Ketamine + ECT; Comparison between the Etomidate + ECT and Ketamine + ECT groups for the recovery rate of Digital Symbol Substitution Task (DSST) reaction time; Test type: Other; p = 0.031, Wilcoxon Signed-Ranked Test — Not adjusted for multiple comparisons
Statistical Analysis 4: Comparison: Ketamine + ECT vs Ketamine Alone; Comparison between the Ketamine + ECT and Ketamine Alone groups for the recovery rate of Digital Symbol Substitution Task (DSST) reaction time; Test type: Other; p = 0.203, Wilcoxon Signed-Ranked Test — Not adjusted for multiple comparisons
Statistical Analysis 5: Comparison: Etomidate + ECT vs Ketamine + ECT; Comparison between the Etomidate + ECT and Ketamine + ECT groups for the recovery rate of Motor Praxis Task (MP) reaction time; Test type: Other; p = 0.008, Wilcoxon Signed-Ranked Test — Not adjusted for multiple comparisons
Statistical Analysis 6: Comparison: Ketamine + ECT vs Ketamine Alone; Comparison between the Ketamine + ECT and Ketamine Alone groups for the recovery rate of Motor Praxis Task (MP) reaction time; Test type: Other; p = 0.496, Wilcoxon Signed-Ranked Test — Not adjusted for multiple comparisons
Statistical Analysis 7: Comparison: Etomidate + ECT vs Ketamine + ECT; Comparison between the Etomidate + ECT and Ketamine + ECT groups for the recovery rate of Visual Object Learning Task (VOLT) reaction time; Test type: Other; p = 0.844, Wilcoxon Signed-Ranked Test — Not adjusted for multiple comparisons
Statistical Analysis 8: Comparison: Ketamine + ECT vs Ketamine Alone; Comparison between the Ketamine + ECT and Ketamine Alone groups for the recovery rate of Visual Object Learning Task (VOLT) reaction time; Test type: Other; p = 0.016, Wilcoxon Signed-Ranked Test — Not adjusted for multiple comparisons
Statistical Analysis 9: Comparison: Etomidate + ECT vs Ketamine + ECT; Comparison between the Etomidate + ECT and Ketamine + ECT groups for the recovery rate of Abstract Matching task (AM) reaction time; Test type: Other; p = 0.062, Wilcoxon Signed-Ranked Test — Not adjusted for multiple comparisons
Statistical Analysis 10: Comparison: Ketamine + ECT vs Ketamine Alone; Comparison between the Ketamine + ECT and Ketamine Alone groups for the recovery rate of Abstract Matching task (AM) reaction time; Test type: Other; p = 0.039, Wilcoxon Signed-Ranked Test — Not adjusted for multiple comparisons

2. Primary Outcome: Change in Cognitive Function During Recovery: Initial Decrement
Description: A cognitive test battery was administered at 0, 30, 60, 90, and 120 minutes following return of consciousness after general anesthesia on each treatment day (1-6). The data from each treatment day (1-6) were averaged for analyses.
  Cognition Test Battery:
  * Psychomotor Vigilance Task (PVT)
  * Digital Symbol Substitution Task (DSST)
  * Motor Praxis Task (MP)
  * Visual Object Learning Task (VOLT)
  * Abstract Matching (AM)
  Initial Decrement for this measure is defined as the difference between response times (in seconds) at baseline and t=0 for each task.
Time Frame: 0, 30, 60, 90, 120 minutes following return of consciousness, assessed on treatment days 1-6.
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | Etomidate + ECT | Ketamine + ECT | Ketamine Alone
Number analyzed (Participants) | 9 | 9 | 11
seconds
  PVT Initial Decrement: number analyzed (Participants) | 7 | 9 | 11
  PVT Initial Decrement | 0.4 [0.4 to 0.4] | 3.5 [2.4 to 5.7] | 6.8 [1.3 to 8.2]
  DSST Initial Decrement: number analyzed (Participants) | 8 | 9 | 11
  DSST Initial Decrement | 2.4 [1.3 to 3.3] | 5.1 [2.7 to 9.3] | 3.1 [2.3 to 12.6]
  MP Initial Decrement | 1.9 [0.6 to 2.8] | 3.0 [1.7 to 4.1] | 2.4 [1.2 to 4.4]
  VOLT Initial Decrement: number analyzed (Participants) | 9 | 7 | 11
  VOLT Initial Decrement | 4.9 [1.4 to 6.6] | 20.9 [20.4 to 21.2] | 6.5 [0.3 to 11.4]
  AM Initial Decrement | 3.2 [1.5 to 4.9] | 2.0 [1.1 to 4.6] | 6.7 [3.2 to 7.8]
Statistical Analysis 1: Comparison: Etomidate + ECT vs Ketamine + ECT; Comparison between the Etomidate + ECT and Ketamine + ECT groups for the initial decrement of Psychomotor Vigilance Task (PVT) reaction time; Test type: Other; p = 0.016, Wilcoxon Signed-Ranked Test — Not adjusted for multiple comparisons
Statistical Analysis 2: Comparison: Ketamine + ECT vs Ketamine Alone; [analysis description as in outcome 1, analysis 2]; Test type: Other; p = 0.039, Wilcoxon Signed-Ranked Test — Not adjusted for multiple comparisons
Statistical Analysis 3: Comparison: Etomidate + ECT vs Ketamine + ECT; Comparison between the Etomidate + ECT and Ketamine + ECT groups for the initial decrement of Digital Symbol Substitution Task (DSST) reaction time; Test type: Other; p = 0.031, Wilcoxon Signed-Ranked Test — Not adjusted for multiple comparisons
Statistical Analysis 4: Comparison: Ketamine + ECT vs Ketamine Alone; Comparison between the Ketamine + ECT and Ketamine Alone groups for the initial decrement of Digital Symbol Substitution Task (DSST) reaction time; Test type: Other; p = 1.0, Wilcoxon Signed-Ranked Test — Not adjusted for multiple comparisons
Statistical Analysis 5: Comparison: Etomidate + ECT vs Ketamine + ECT; Comparison between the Etomidate + ECT and Ketamine + ECT groups for the initial decrement of Motor Praxis task (MP) reaction time; Test type: Other; p = 0.195, Wilcoxon Signed-Ranked Test — Not adjusted for multiple comparisons
Statistical Analysis 6: Comparison: Ketamine + ECT vs Ketamine Alone; Comparison between the Ketamine + ECT and Ketamine Alone groups for the initial decrement of Motor Praxis task (MP) reaction time; Test type: Other; p = 0.570, Wilcoxon Signed-Ranked Test — Not adjusted for multiple comparisons
Statistical Analysis 7: Comparison: Etomidate + ECT vs Ketamine + ECT; Comparison between the Etomidate + ECT and Ketamine + ECT groups for the initial decrement of Visual Object Learning Task (VOLT) reaction time; Test type: Other; p = 0.031, Wilcoxon Signed-Ranked Test — Not adjusted for multiple comparisons
Statistical Analysis 8: Comparison: Ketamine + ECT vs Ketamine Alone; Comparison between the Ketamine + ECT and Ketamine Alone groups for the initial decrement of Visual Object Learning Task (VOLT) reaction time; Test type: Other; p = 0.016, Wilcoxon Signed-Ranked Test — Not adjusted for multiple comparisons
Statistical Analysis 9: Comparison: Etomidate + ECT vs Ketamine + ECT; Comparison between the Etomidate + ECT and Ketamine + ECT groups for the initial decrement of Abstract Matching (AM) task reaction time; Test type: Other; p = 1.00, Wilcoxon Signed-Ranked Test — Not adjusted for multiple comparisons
Statistical Analysis 10: Comparison: Ketamine + ECT vs Ketamine Alone; Comparison between the Ketamine + ECT and Ketamine Alone groups for the initial decrement of Abstract Matching (AM) task reaction time; Test type: Other; p = 0.109, Wilcoxon Signed-Ranked Test — Not adjusted for multiple comparisons

3. Secondary Outcome: Delirium Incidence and Severity
Description: Assessed using 3D Confusion Assessment Method (CAM).
  The groups/arms for this outcome are separated by anesthetic regimen; however, due to the crossover design of this study all participants are included in analyses for each group.
Time Frame: Immediately following return of consciousness (t=0) during treatment days 1-6.
Population: All participants (12) who completed both baseline and t=0 delirium assessments on at least one treatment day.
Measure: Number; unit: Delirium Assessments
Units Other Than Participants: Delirium Assessments
Arm/Group | Ketamine + ECT | Etomidate + ECT | Ketamine Alone
Number analyzed (Participants) | 12 | 12 | 12
Number analyzed (Delirium Assessments) | 42 | 46 | 44
Delirium Assessments
  Positive Delirium at Baseline | 1 | 0 | 0
  Negative Delirium at Baseline | 20 | 23 | 23
  Positive Delirium at t=0 | 1 | 0 | 2
  Negative Delirium at t=0 | 20 | 23 | 19

4. Secondary Outcome: Suicidality
Description: The groups/arms for this outcome are combined as a whole-group analysis due to the crossover design of this study, as pre-specified by the study protocol. Breaking up the analyses into the various arms of the study would change our scientific questions and approach. All participants included in analyses completed all treatments, the various arms for the study vary only in the order in which participants received each treatment. These data show the change in suicidality from baseline to treatment 6 based on the Scale of Suicide Ideation.
  The measure completed was the Scale of Suicide Ideation. For this study, participants completed the following questions of the questionnaire:
  1. wish to live (0 Moderate to Strong, 1 Weak, 2 None)
  2. wish to die (0 None, 1 Weak, 2 Moderate to Strong)
  The total scores range from 0-4. Lower scores indicate high suicide ideation, and high scores indicate low suicide ideation.
Time Frame: assessed at baseline on treatment days 1-6.
Population: 114 Assessments of suicidality were completed across 13 participants on days 1-6. Data reported show the average change in suicidality from baseline to treatment 6 based on the Scale of Suicide Ideation.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Suicide Assessments
Groups:
- All Participants: All participants enrolled in study procedures
Arm/Group | All Participants
Number analyzed (Participants) | 13
Number analyzed (Suicide Assessments) | 114
score on a scale
  Change in Will to live | 0.077 (0.277)
  Change in Will to die | 0.077 (0.277)

5. Secondary Outcome: ECT Seizure Duration
Description: Duration (in seconds) of seizure induced by ECT treatment
Time Frame: up to days 1-6
Population: These data were not collected from patient ECT procedure records and therefore were not analyzed.
Arm/Group | All Participants
Number analyzed (Participants) | 0

6. Secondary Outcome: ECT Electrical Dose
Description: The electrical dose necessary for seizure induction is determined during a dose-charge titration session prior to participant randomization and session 1. These results report the average electrical dose across all participants for the first treatment session during Treatment Week 1.
  The range for these data is 0 - 100% electrical charge.
Time Frame: First ECT treatment session during Treatment Week 1
Population: Results are shown for all 13 participants who completed at least one treatment session following the dose charge titration session.
Measure: Mean (Standard Deviation); unit: percentage of electrical charge
Arm/Group | All Participants
Number analyzed (Participants) | 13
percentage of electrical charge | 32.5 (8.66)

7. Secondary Outcome: Subjective Assessment of Whether ECT Was Performed, Determined by Asking the Patient.
Description: To assess patient blinding of treatment performed, the patient will be asked: "Based on how you feel, did you have ECT today?"
  Results indicate participants correctly answering the subjective assessment.
Time Frame: Assessed at 120 minutes after return of responsiveness on treatment days 1-6
Population: The sample analyzed for each group consists of the total number of treatments performed with paired subjective assessments out of 12 participants.
Measure: Count of Units; unit: Subjective Assessments w/ paired Tx
Units Other Than Participants: Subjective Assessments w/ paired Tx
Arm/Group | Etomidate + ECT | Ketamine + ECT | Ketamine Alone
Number analyzed (Participants) | 12 | 12 | 12
Number analyzed (Subjective Assessments w/ paired Tx) | 23 | 21 | 22
Subjective Assessments w/ paired Tx | 18 | 18 | 6

8. Secondary Outcome: Change in Mood Assessed Using the Mood Self-Assessment Manikin
Description: Mood Self-Assessment Manikin (SAM) Scale: 1 (very unpleasant) - 9 (very pleasant).
  The groups/arms for this outcome are combined as a whole-group analysis due to the Crossover design of this study, as pre-specified by the study protocol. Breaking up the analyses into the various arms of the study would change our scientific questions and approach. Further, any statistical analyses would be underpowered due to low participant numbers in each arm. Thus, the results are combined and reported as a whole group analysis. All participants included in analyses completed all treatments included in the study, the various arms for the study vary only in the order in which participants received each treatment. These data show the change in mood from baseline to treatment 6 based on the SAM. Additionally, data collected at baseline are not dependent on the study group/arm.
Time Frame: baseline and 120 minutes after return of responsiveness, assessed on treatment days 1-6
Population: The average change in SAM score from baseline to t=120 for all sessions across all participants (t=120 - baseline).
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: SAM Assessments
Arm/Group | AllParticipants
Number analyzed (Participants) | 13
Number analyzed (SAM Assessments) | 64
score on a scale | -0.266 (1.043)

9. Secondary Outcome: Average Change in Mood Based on the Depression PROMIS-CAT
Description: PROMIS-CAT (Patient Reported Outcomes Measurement Information System-Computer Adaptive Testing) for depression
  The groups/arms for this outcome are combined as a whole-group analysis due to the Crossover design of this study, as pre-specified by the study protocol. Breaking up the analyses into the various arms of the study would change our scientific questions and approach. Further, any statistical analyses would be underpowered due to low participant numbers in each arm. Thus, the results are combined and reported as a whole group analysis. All participants included in analyses completed all treatments included in the study, the various arms for the study vary only in the order in which participants received each treatment. These data show the change in mood from baseline to treatment 6 based on the PROMIS-CAT. Additionally, data collected at baseline are not dependent on the study group/arm.
Time Frame: baseline and 120 minutes after return of responsiveness, assessed on treatment days 1-6
Population: All 13 participants who completed the depression PROMS-CAT both before and after treatment (baseline and 120 minutes following return of responsiveness) on at least one treatment day.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 13
score on a scale | -0.5108 (1.975)

10. Secondary Outcome: Change in Delta Band (0.5-4 Hz) Relative Power in the Scale EEG During Recovery
Description: High-density EEG collected during 5-minute epochs of eyes-closed quiet resting at baseline and post-ECT. Results are reported as the percent of total power in the delta band over the sum of total power between 0.5 - 70Hz.
Time Frame: baseline, post-ECT from 0-120 minutes
Population: Participants with EEG data collected at baseline at T0 post-ECT for at least 1 ECT session were included in analyses.
Measure: Median (Inter-Quartile Range); unit: percent of total power
Arm/Group | Etomidate + ECT | Ketamine + ECT | Ketamine Alone
Number analyzed (Participants) | 9 | 9 | 10
percent of total power | -0.064 [-0.182 to 0.033] | -0.111 [-0.160 to 0.00] | -0.038 [-0.106 to 0.118]
Statistical Analysis 1: Comparison: Etomidate + ECT; Comparison of relative power in the delta band at baseline compared to T0 following return of responsiveness; Test type: Other; p = 0.301, Wilcoxon signed-rank paired test
Statistical Analysis 2: Comparison: Ketamine + ECT; Comparison of relative power in the delta band at baseline compared to T0 following return of responsiveness; Test type: Other; p = 0.301, Wilcoxon signed-rank paired test
Statistical Analysis 3: Comparison: Ketamine Alone; Comparison of relative power in the delta band at baseline compared to T0 following return of responsiveness; Test type: Other; p = 0.557, Wilcoxon signed-rank paired test

11. Secondary Outcome: Change in Theta Band (4-8 Hz) Relative Power in the Scalp EEG During Recovery
Description: High-density EEG collected during 5-minute epochs of eyes-closed quiet resting at baseline and post-ECT. Results are reported as the percent of total power in the theta band over the sum of total power between 0.5 - 70Hz.
Time Frame: baseline, post-ECT from 0-120 minutes
Population: Participants with EEG data collected at baseline at T0 post-ECT for at least 1 ECT session were included in analyses.
Measure: Median (Inter-Quartile Range); unit: percent of total power
Arm/Group | Etomidate + ECT | Ketamine + ECT | Ketamine Alone
Number analyzed (Participants) | 9 | 9 | 10
percent of total power | -0.008 [-0.048 to 0.051] | -0.015 [-0.038 to 0.077] | 0.015 [-0.040 to 0.156]
Statistical Analysis 1: Comparison: Etomidate + ECT; Comparison of relative power in the theta band at baseline compared to T0 following return of responsiveness; Test type: Other; p = 0.910, Wilcoxon signed-rank paired test
Statistical Analysis 2: Comparison: Ketamine + ECT; Comparison of relative power in the theta band at baseline compared to T0 following return of responsiveness; Test type: Other; p = 0.734, Wilcoxon signed-rank paired test
Statistical Analysis 3: Comparison: Ketamine Alone; Comparison of relative power in the theta band at baseline compared to T0 following return of responsiveness; Test type: Other; p = 0.322, Wilcoxon signed-rank paired test

12. Secondary Outcome: Change in Alpha Band (8-13 Hz) Power in the Scalp EEG During Recovery
Description: High-density EEG collected during 5-minute epochs of eyes-closed quiet resting at baseline and post-ECT. Results are reported as the percent of total power in the alpha band over the sum of total power between 0.5 - 70Hz.
Time Frame: baseline, post-ECT from 0-120 minutes
Population: Participants with EEG data collected at baseline at T0 post-ECT for at least 1 ECT session were included in analyses.
Measure: Median (Inter-Quartile Range); unit: percent of total power
Arm/Group | Etomidate + ECT | Ketamine + ECT | Ketamine Alone
Number analyzed (Participants) | 9 | 9 | 10
percent of total power | 0.016 [-0.001 to 0.142] | 0.053 [0.016 to 0.112] | 0.006 [-0.026 to 0.053]
Statistical Analysis 1: Comparison: Etomidate + ECT; Comparison of relative power in the alpha band at baseline compared to T0 following return of responsiveness; Test type: Other; p = 0.164, Wilcoxon signed-rank paired test
Statistical Analysis 2: Comparison: Ketamine + ECT; Comparison of relative power in the alpha band at baseline compared to T0 following return of responsiveness; Test type: Other; p = 0.039, Wilcoxon signed-rank paired test
Statistical Analysis 3: Comparison: Ketamine Alone; Comparison of relative power in the alpha band at baseline compared to T0 following return of responsiveness; Test type: Other; p = 0.375, Wilcoxon signed-rank paired test

13. Secondary Outcome: Change in Beta Band (13-20 Hz) Relative Power in the Scalp EEG During Recovery
Description: High-density EEG collected during 5-minute epochs of eyes-closed quiet resting at baseline and post-ECT. Results are reported as the percent of total power in the beta band over the sum of total power between 0.5 - 70Hz.
Time Frame: baseline, post-ECT from 0-120 minutes
Population: Participants with EEG data collected at baseline at T0 post-ECT for at least 1 ECT session were included in analyses.
Measure: Median (Inter-Quartile Range); unit: percent of total power
Arm/Group | Etomidate + ECT | Ketamine + ECT | Ketamine Alone
Number analyzed (Participants) | 9 | 9 | 10
percent of total power | -0.001 [-0.010 to 0.029] | -0.004 [-0.012 to 0.039] | -0.008 [-0.019 to 0.014]
Statistical Analysis 1: Comparison: Etomidate + ECT; Comparison of relative power in the beta band at baseline compared to T0 following return of responsiveness; Test type: Other; p = 0.910, Wilcoxon signed-rank paired test
Statistical Analysis 2: Comparison: Ketamine + ECT; Comparison of relative power in the beta band at baseline compared to T0 following return of responsiveness; Test type: Other; p = 0.910, Wilcoxon signed-rank paired test
Statistical Analysis 3: Comparison: Ketamine Alone; Comparison of relative power in the beta band at baseline compared to T0 following return of responsiveness; Test type: Other; p = 0.625, Wilcoxon signed-rank paired test

14. Secondary Outcome: Change in Anterior-Posterior Functional Connectivity in the Scalp During Recovery
Description: High-density EEG collected during 5-minute epochs of eyes-closed quiet resting at baseline and post-ECT. Results are reported as the coherence measure, which is used for tracking changes in anterior-posterior functional connectivity.
  Coherence is a measure of synchronization between two signals which is used to measure anterior-posterior functional connectivity. Coherence is a unitless measure between 0 and 1. High coherence between time-series of two neural populations reflects higher efficiency in communication between those populations and therefore stronger functional connectivity.
Time Frame: baseline, post-ECT from 0-120 minutes
Population: Participants with EEG data collected at baseline at T0 post-ECT for at least 1 ECT session were included in analyses.
Measure: Median (Inter-Quartile Range); unit: unitless
Arm/Group | Etomidate + ECT | Ketamine + ECT | Ketamine Alone
Number analyzed (Participants) | 9 | 9 | 10
unitless | -0.014 [-0.052 to 0.004] | -0.002 [-0.010 to 0.014] | -0.004 [-0.043 to 0.0023]
Statistical Analysis 1: Comparison: Etomidate + ECT; Comparison of anterior-posterior functional connectivity (coherence) at baseline compared to T0 following return of responsiveness; Test type: Other; p = 0.129, Wilcoxon signed-rank paired test
Statistical Analysis 2: Comparison: Ketamine + ECT; [analysis description as in outcome 14, analysis 1]; Test type: Other; p = 0.910, Wilcoxon signed-rank paired test
Statistical Analysis 3: Comparison: Ketamine Alone; [analysis description as in outcome 14, analysis 1]; Test type: Other; p = 0.625, Wilcoxon signed-rank paired test

15. Secondary Outcome: Change in Anterior-Posterior Phase-lag in the Scalp EEG During Recovery
Description: High-density EEG collected during 5-minute epochs of eyes-closed quiet resting at baseline and post-ECT. Phase-lag was assessed using the Phase-Lag Index (PLI), a measure ranging from 0 - 1. A consistent phase-lag between two tim-series results in a PLI of 1. A time-series without coupling results in a PLI near or equaling 0. Results show the difference in anterior-posterior PLI between baseline and post-ECT.
Time Frame: baseline, post-ECT from 0 -120 minutes
Measure: Median (Inter-Quartile Range); unit: Phase Lag Index (PLI)
Arm/Group | Etomidate + ECT | Ketamine + ECT | Ketamine Alone
Number analyzed (Participants) | 9 | 9 | 10
Phase Lag Index (PLI) | -0.001 [-0.034 to 0.044] | -0.049 [-0.089 to 0.066] | -0.017 [-0.058 to -0.005]
Statistical Analysis 1: Comparison: Etomidate + ECT; Comparison of anterior-posterior phase-lag (PLI) at baseline compared to T0 following return of responsiveness; Test type: Other; p = 1.000, Wilcoxon signed-rank paired test
Statistical Analysis 2: Comparison: Ketamine + ECT; Comparison of anterior-posterior phase-lag (PLI) at baseline compared to T0 following return of responsiveness; Test type: Other; p = 0.496, Wilcoxon signed-rank paired test
Statistical Analysis 3: Comparison: Ketamine Alone; Comparison of anterior-posterior phase-lag (PLI) at baseline compared to T0 following return of responsiveness; Test type: Other; p = 0.160, Wilcoxon signed-rank paired test

16. Secondary Outcome: Change in EEG Entropy in the Scalp EEG During Recovery
Description: High-density EEG collected during 5-minute epochs of eyes-closed quiet resting at baseline and post-ECT. Results are reported as permutation entropy (PE) measures in posterior regions, which we are using to track changes in scalp EEG entropy.
  Permutation Entropy (PE) is a measure that is used to quantify the complexity of time series signals. It is a unitless measure between 0 and 1. Lower the PE represents a more regular and more deterministic time series while higher PE represents a more complex time series.
Time Frame: baseline, Post-ECT from 0 -120 minutes
Population: Participants with EEG data collected at baseline at T0 post-ECT for at least 1 ECT session were included in analyses.
Measure: Median (Inter-Quartile Range); unit: unitless
Arm/Group | Etomidate + ECT | Ketamine + ECT | Ketamine Alone
Number analyzed (Participants) | 9 | 9 | 10
unitless | -0.018 [-0.047 to -0.005] | -0.003 [-0.039 to 0.013] | -0.006 [-0.012 to 0.003]
Statistical Analysis 1: Comparison: Etomidate + ECT; Comparison of EEG Entropy using Permutation Entropy (PE) measures at baseline compared to T0 following return of responsiveness; Test type: Other; p = 0.008, Wilcoxon Signed-Ranked Test
Statistical Analysis 2: Comparison: Ketamine + ECT; [analysis description as in outcome 16, analysis 1]; Test type: Other; p = 0.359, Wilcoxon Signed-Ranked Test
Statistical Analysis 3: Comparison: Ketamine Alone; [analysis description as in outcome 16, analysis 1]; Test type: Other; p = 0.375, Wilcoxon Signed-Ranked Test

ADVERSE EVENTS:
Time Frame: approximately 3 weeks
Description: Each group/arm of this crossover study were reported separately. All participants who completed at least 1 treatment session were included in adverse event reporting.
  Each group contains a total of 15 participants, as each participant completed each arm of the study at least once.
Groups:
- Ketamine +ECT: General anesthesia for ECT will be induced with ketamine, approximately 2 mg/kg (1-2.5 mg/kg). Following application of stimulation electrodes to the patients scalp, an ECT charge will be administered at the previously determined therapeutic dose.
- Etomidate +ECT: General anesthesia for ECT will be induced with etomidate, approximately 0.2 mg/kg (0.1-0.6 mg/kg). Following application of stimulation electrodes to the patients scalp, an ECT charge will be administered at the previously determined therapeutic dose.
- Ketamine Sham: General anesthesia for ECT will be induced with ketamine, approximately 2 mg/kg (1-2.5 mg/kg). Following application of stimulation electrodes to the patients scalp, no ECT charge will be administered.
Arm/Group | Ketamine +ECT | Etomidate +ECT | Ketamine Sham
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-25): https://cdn.clinicaltrials.gov/large-docs/30/NCT02761330/Prot_SAP_000.pdf